The Effectiveness of Fixed Dose Combination of Alpha Lipoic Acid and Vitamin B Preparation for Treatment of Diabetic Polyneuropathy in Type 2 diabetes mellitus patients: A randomized placebo-controlled trial.

**DATE: 31ST MARCH 2024** 

| APPENDIX I: Case report form | <b>DATE</b> : | ID: |
|------------------------------|---------------|-----|
| Name: | | |
| IC: | | |
| RN: | | |

#### A. BASELINE VISIT

Research topic: The Effectiveness of Fixed Dose Combination of Alpha Lipoic Acid and Vitamin B Preparations for Treatment of Diabetic Polyneuropathy in Type 2 diabetes mellitus patients: A randomized placebo-controlled trial

#### **SECTION A:**

SCREENING CRITERIA FOR ELIGIBILITY TO PARTICIPATE IN THE STUDY USING NEUROLOGICAL SYMPTOM SCORE (NSS) AND NEUROPATHY DISABILITY SCORE (NDS) QUESTIONS

(Questions and examination of diabetic polyneuropathy will be done by trained research supervisors)

Neuropathy Symptom Score (NSS) and Neuropathy Disability Score (NDS)

| Symptoms | |
|-------------------------------------|---|
| Burning, numbness, tingling | 2 |
| Fatigue, cramping, aching | 1 |
| None | 0 |
| Location | |
| Feet | 2 |
| Calves | 1 |
| Elsewhere | 0 |
| Timing of symptoms | |
| Nocturnal exacerbation | 2 |
| Present during day and night | 1 |
| Present during the day only | 0 |
| Symptoms wake patient up from sleep | 1 |
| Manoeuvres to reduce symptoms | |
| Walking | 2 |
| Standing | 1 |
| Sitting/Lying | 0 |
| NSS score | |

| Absent/reduced 1 1 1 Present 0 0 0 Temperature (tip of cold tuning fork at dorsum of the footabove medial malleolus) Absent/reduced 1 1 1 Present 0 0 0 Pin-prick (apply pin at proximal end of big toenail to distinguish sharp/blunt) Absent/reduced 1 1 1 Present 0 0 0 Ankle reflex Absent Absent 2 2 2 Present only with re-enforcement 1 1 Present 1 0 0 | Signs | Right | Left |
|---|---|---|---|
| Present 0 0 Temperature (tip of cold tuning fork at dorsum of the footabove medial malleolus) Absent/reduced 1 1 Present 0 0 Pin-prick (apply pin at proximal end of big toenail to distinguish sharp/blunt) Absent/reduced 1 1 Present 0 0 0 Ankle reflex Absent 2 2 Present only with re-enforcement 1 1 | Vibration (128 Hz turning fork at the hallux of the big toe) | | |
| Present 0 0 Temperature (tip of cold tuning fork at dorsum of the footabove medial malleolus) Absent/reduced 1 1 Present 0 0 Pin-prick (apply pin at proximal end of big toenail to distinguish sharp/blunt) Absent/reduced 1 1 Present 0 0 0 Ankle reflex Absent 2 2 Present only with re-enforcement 1 1 | | | |
| Absent/reduced 1 1 1 Present 0 0 0 Pin-prick (apply pin at proximal end of big toenail to distinguish sharp/blunt) Absent/reduced 1 1 1 Present 0 0 0 Ankle reflex Absent 2 2 2 Present only with re-enforcement 1 1 | Absent/reduced | 1 | 1 |
| Absent/reduced 1 1 1 Present 0 0 0 Pin-prick (apply pin at proximal end of big toenail to distinguish sharp/blunt) Absent/reduced 1 1 1 Present 0 0 0 Ankle reflex Absent 2 2 2 Present only with re-enforcement 1 1 | Present | 0 | 0 |
| Present 0 0 0 Pin-prick (apply pin at proximal end of big toenail to distinguish sharp/blunt) Absent/reduced 1 1 1 Present 0 0 0 Ankle reflex Absent 2 2 2 Present only with re-enforcement 1 1 | | | |
| Present 0 0 0 Pin-prick (apply pin at proximal end of big toenail to distinguish sharp/blunt) Absent/reduced 1 1 1 Present 0 0 0 Ankle reflex Absent 2 2 2 Present only with re-enforcement 1 1 | | | |
| Pin-prick (apply pin at proximal end of big toenail to distinguish sharp/blunt) Absent/reduced Present O Ankle reflex Absent Present 0 2 2 Present only with re-enforcement 1 | Absent/reduced | 1 | 1 |
| Absent/reduced 1 1 Present 0 0 Ankle reflex 2 2 Present only with re-enforcement 1 1 | Present | 0 | 0 |
| Present 0 0 Ankle reflex 2 2 Absent 2 2 Present only with re-enforcement 1 1 | | | |
| Ankle reflex Absent 2 2 Present only with re-enforcement 1 1 | Absent/reduced | 1 | 1 |
| Absent 2 2 Present only with re-enforcement 1 1 | | 0 | 0 |
| Present only with re-enforcement 1 1 | | | |
| | | 2 | |
| Precent | , and the second | 1 | |
| Total NDS | | U | U |

Symptoms: Mild (NSS 3-4), Moderate (NSS 5-6), Severe (NSS 7-9)

Signs: Mild (NDS 3-5), Moderate (NDS 6-8), Severe (9-10)

#### The minimum acceptable criteria for a diagnosis of peripheral neuropathy were:

- 1. Presence of moderate signs (NDS >6) regardless of symptoms OR
- 2. Mild signs (NDS > 3) with moderate symptoms (NSS > 5)

#### **SECTION B**

Research topic: The Effectiveness of Fixed Dose Combination of Alpha Lipoic Acid and Vitamin B Preparations for Treatment of Diabetic Polyneuropathy in Type 2 diabetes mellitus patients: A randomized placebo-controlled trial

#### **B1: PARTICIPANT BACKGROUND**

| 1. | Gender | □ Male | □ Female |
|-----|--------------------|-----------------------|----------|
| 2. | Age | | |
| 3. | Race | □ Malay | |
| | | □ Chinese | |
| | | □ Indian | |
| | | □ Siamese | |
| | | □ Others | |
| | | Please state | |
| 4. | Level of Education | □ Not going to school | 1 |
| | | ☐ Elementary School | |
| | | □ High School | |
| | | □ University | |
| 5. | Jobs | □ Working | |
| | | □ Not Working | |
| 6. | Monthly income | | |
| | - | RM | |
| 7. | Marriage status | □ Single | |
| / . | Trainingo status | □ Married | |
| | | L Mullion | |

# **B2: HEALTH INFORMATION AND DIABETES INFORMATION** (To be filled in by the researcher)

| 1. | How long have you had diabetes? | |
|----|-----------------------------------|-------------------------|
| | | Years |
| 2. | Diabetes medication | □ Metformin |
| | | □ Gliclazide |
| | | □ SGLT-2 |
| | | □ DPP4 inhibitor |
| | | □ Insulin |
| | | □ Others: Please state: |
| 4. | Do you have high blood pressure? | □ Yes |
| | | □ No |
| 5. | Do you have high cholesterol? | □Yes |
| | | □ No |
| 6. | Retinopathy | □Yes |
| | | □ No |
| 7. | Ischemic Heart Disease/Myocardial | □Yes |
| | Infarction | □ No |
| 8. | Other diseases: | |
| | Specify | |
| 9. | History of allergy to medication | □ Yes |
| | | □ No |

## **B3:** Total symptoms score (TSS)

| Neuropathic | Symptoms frequency | | Symptom intensity | | |
|---|---|---|---|---|---|
| symptoms | | Absent | Slight | Moderate | Severe |
| 1. Stabbing | Occasional | 0 | 1.00 | 2.00 | 3.00 |
| Pain | Frequent | 0 | 1.33 | 2.33 | 3.33 |
| | Almost continues | 0 | 1.66 | 2.66 | 3.66 |

| Neuropathic | Symptoms frequency | | Symptom intensity | | |
|---|---|---|---|---|---|
| symptoms | | Absent Slight Moderate | | | |
| 2.Burning | Occasional | 0 | 1.00 | 2.00 | 3.00 |
| pain | Frequent | 0 | 1.33 | 2.33 | 3.33 |
| | Almost continues | 0 | 1.66 | 2.66 | 3.66 |

| Neuropathic | Symptoms frequency | Symptom intensity | | | |
|---|---|---|---|---|---|
| symptoms | | Absent | Slight | Moderate | Severe |
| 3.Paraesthesia | Occasional | 0 | 1.00 | 2.00 | 3.00 |
| | Frequent | 0 | 1.33 | 2.33 | 3.33 |
| | Almost continues | 0 | 1.66 | 2.66 | 3.66 |

| Neuropathic | Symptoms frequency | | Symptom intensity | | |
|---|---|---|---|---|---|
| symptoms | | Absent | Severe | | |
| 4.Numbness | Occasional | 0 | 1.00 | 2.00 | 3.00 |
| | Frequent | 0 | 1.33 | 2.33 | 3.33 |
| | Almost continues | 0 | 1.66 | 2.66 | 3.66 |

| Symptom frequency | Sympton | n intensit | y | |
|---------------------|---------|------------|----------|--------|
| | Absent | Slight | Moderate | Severe |
| Occasional | 0 | 1.00 | 2.00 | 3.00 |
| Frequent | 0 | 1.33 | 2.33 | 3.33 |
| (Almost) continuous | 0 | 1.66 | 2.66 | 3.66 |

## B4: The revised version of Diabetes Quality of Life (RV-DQoL) questionnaire

Please read each statement carefully and mark the number that best suits you.

| Satisfaction Domain | Very satisfied | Moderately satisfied | Neither<br>satisfied nor<br>dissatisfied | Moderately<br>dissatisfied | Very<br>dissatisfied |
|---|---|---|---|---|---|
| How satisfied are you with the amount of time it takes to manage your diabetes? | 1 | 2 | 3 | 4 | 5 |
| 2. How satisfied are you with the amount of time you spend getting checkups? | 1 | 2 | 3 | 4 | 5 |
| 3. How satisfied are you with the time it takes to determine your sugar level? | 1 | 2 | 3 | 4 | 5 |
| 4. How satisfied are you with your current treatment? | 1 | 2 | 3 | 4 | 5 |

| 5. How satisfied are you with your knowledge about your diabetes? | 1 | 2 | 3 | 4 | 5 |
|---|---|---|---|---|---|
| 6. How satisfied are you with life in general? | 1 | 2 | 3 | 4 | 5 |

| Impact Domain | Never | Sometimes | Often | Frequently | Always |
|---|---|---|---|---|---|
| How often do you feel pain associated with the treatment for your diabetes? | 1 | 2 | 3 | 4 | 5 |
| 2. How often do you feel physically ill? | 1 | 2 | 3 | 4 | 5 |
| 3. How often does your diabetes interfere with your family life? | 1 | 2 | 3 | 4 | 5 |
| 4. How often do you find your diabetes limiting your social relationships and friendships? | 1 | 2 | 3 | 4 | 5 |

| Worry Domain | Never | Sometimes | Often | Frequently | Always |
|---|---|---|---|---|---|
| 1. How often do you worry about whether you will pass out? | 1 | 2 | 3 | 4 | 5 |
| 2. How often do you worry that your body looks different because you have diabetes? | 1 | 2 | 3 | 4 | 5 |
| 3. How often do your worry that you will get complications from your diabetes? | 1 | 2 | 3 | 4 | 5 |

## **B5:** Clinical data

| 1 | body mass index (BMI) | kg/m <sup>2</sup> |
|---|-----------------------|-------------------|
| | Weight: | |
| | Height: | |
| 2 | Blood Pressure | |
| | | mmHg |

### **B6:** Blood test results at the first visit

| Blood Test | Result |
|--------------|--------|
| FBS (mmol/L) | |
| Hba1c (%) | |
| TC (mmol/L) | |
| LDL (mmol/L) | |
| HDL (mmol/L) | |
| TG (mmol/L) | |
| Creatinine | |
| Urea | |
| AST | |
| ALT | |
| ALP | |

| B. SECOND VISIT | (6 WEEKS) | <b>DATE</b> : | ID: |
|-----------------|-----------|---------------|-----|

Research topic: The Effectiveness of Fixed Dose Combination of Alpha Lipoic Acid and Vitamin B Preparations for Treatment of Diabetic Polyneuropathy in Type 2 diabetes mellitus patients: A randomized placebo-controlled trial

| Name: | <br> |
|-------|------|
| IC: | |
| RN: | |

# 1. Total symptoms score (TSS)

| Neuropathic | Symptoms frequency | Symptom intensity | | | |
|---|---|---|---|---|---|
| symptoms | | Absent | Slight | Moderate | Severe |
| 1. Stabbing | Occasional | 0 | 1.00 | 2.00 | 3.00 |
| Pain | Frequent | 0 | 1.33 | 2.33 | 3.33 |
| | Almost continues | 0 | 1.66 | 2.66 | 3.66 |

| Neuropathic | Symptoms frequency | Symptom intensity | | | |
|---|---|---|---|---|---|
| symptoms | | Absent | Slight | Moderate | Severe |
| 2.Burning | Occasional | 0 | 1.00 | 2.00 | 3.00 |
| pain | Frequent | 0 | 1.33 | 2.33 | 3.33 |
| | Almost continues | 0 | 1.66 | 2.66 | 3.66 |

| Neuropathic | Symptoms frequency | Sympto | Symptom intensity | | |
|---|---|---|---|---|---|
| symptoms | | Absent | Slight | Moderate | Severe |
| 3.Paraesthesia | Occasional | 0 | 1.00 | 2.00 | 3.00 |
| | Frequent | 0 | 1.33 | 2.33 | 3.33 |
| | Almost continues | 0 | 1.66 | 2.66 | 3.66 |

| Neuropathic | Symptoms frequency | Symptom intensity | | | |
|---|---|---|---|---|---|
| symptoms | | Absent | Slight | Moderate | Severe |
| 4.Numbness | Occasional | 0 | 1.00 | 2.00 | 3.00 |
| | Frequent | 0 | 1.33 | 2.33 | 3.33 |
| | Almost continues | 0 | 1.66 | 2.66 | 3.66 |

# 2. Neuropathy Symptom Score (NSS)

| Symptoms | |
|-------------------------------------|---|
| Burning, numbness, tingling | 2 |
| Fatigue, cramping, aching | 1 |
| None | 0 |
| Location | |
| Feet | 2 |
| Calves | 1 |
| Elsewhere | 0 |
| Timing of symptoms | |
| Nocturnal exacerbation | 2 |
| Present during day and night | 1 |
| Present during the day only | 0 |
| Symptoms wake patient up from sleep | 1 |
| Manoeuvres to reduce symptoms | |
| Walking | 2 |
| Standing | 1 |
| Sitting/Lying | 0 |
| NSS score | |

## B4: The revised version of Diabetes Quality of Life (RV-DQoL) questionnaire

Please read each statement carefully and mark the number that best suits you.

| Satisfaction Domain | Very satisfied | Moderately satisfied | Neither<br>satisfied nor<br>dissatisfied | Moderately<br>dissatisfied | Very<br>dissatisfied |
|---|---|---|---|---|---|
| 7. How satisfied are you with the amount of time it takes to manage your diabetes? | 1 | 2 | 3 | 4 | 5 |
| 8. How satisfied are you with the amount of time you spend getting checkups? | 1 | 2 | 3 | 4 | 5 |
| 9. How satisfied are you with the time it takes to determine your sugar level? | 1 | 2 | 3 | 4 | 5 |
| 10. How satisfied are you with your current treatment? | 1 | 2 | 3 | 4 | 5 |

| 11. How satisfied are you with your knowledge about your diabetes? | 1 | 2 | 3 | 4 | 5 |
|---|---|---|---|---|---|
| 12. How satisfied are you with life in general? | 1 | 2 | 3 | 4 | 5 |

| Impact Domain | Never | Sometimes | Often | Frequently | Always |
|---|---|---|---|---|---|
| 5. How often do you feel pain associated with the treatment for your diabetes? | 1 | 2 | 3 | 4 | 5 |
| 6. How often do you feel physically ill? | 1 | 2 | 3 | 4 | 5 |
| 7. How often does your diabetes interfere with your family life? | 1 | 2 | 3 | 4 | 5 |
| 8. How often do you find your diabetes limiting your social relationships and friendships? | 1 | 2 | 3 | 4 | 5 |

| Worry Domain | Never | Sometimes | Often | Frequently | Always |
|---|---|---|---|---|---|
| 4. How often do you worry about whether you will pass out? | 1 | 2 | 3 | 4 | 5 |
| 5. How often do you worry that your body looks different because you have diabetes? | 1 | 2 | 3 | 4 | 5 |
| 6. How often do your worry that you will get complications from your diabetes? | 1 | 2 | 3 | 4 | 5 |

| | . Clinical Data | | |
|---|---|---|---|
| 1 | Body mass index (BMI) | | kg/m <sup>2</sup> |
| | Weight: | | |
| | Height: | | |
| 2 | Blood Pressure | | *** |
| | | | mmHg |
| 1 | . Medication side effect: | | |
| 7 | Yes | $\square$ No | |
| | State if applicable: | | |
| | i | | |
| 5 | . Do you take medicine ev | ery day? | ? |
| | □Yes | □No | |
| 6 | . If you do not take medic medicine? | ine ever | y day, state how often in a week you do not tak |
| | ☐ Once a week | | |
| | $\Box$ 2-3 times a week | | |
| | ☐ More than 3 times a we | eek | |
| 7 | . State the reason you are | not taki | ng medicine |
| | ☐ Forgot | | |
| | ☐ Side effects | _ | |
| | ☐ Others reasons - Specia | fy | |

| C. | 3 <sup>RD</sup> | <b>VISIT</b> | (12 | WEEKS) | ) |
|----|-----------------|--------------|-----|-----------|---|
| • | • | , 1011 | | TT LLIED, | , |

| C. 3 <sup>RD</sup> VISIT (12 WEEKS) | <b>DATE</b> : | ID: |
|---|---|---|
| Research topic: The Effectiveness of Fix | ed Dose Combination of Alpha | a Lipoic Acid and |

Research topic: The Effectiveness of Fixed Dose Combination of Alpha Lipoic Acid and Vitamin B Preparations for Treatment of Diabetic Polyneuropathy in Type 2 diabetes mellitus patients: A randomized placebo-controlled trial

| Name: |
|-------|
| IC: |
| RN: |

#### 1. Total symptoms score (TSS)

| Neuropathic | Symptoms frequency | Symptom intensity | | | |
|---|---|---|---|---|---|
| symptoms | | Absent | Slight | Moderate | Severe |
| 1. Stabbing | Occasional | 0 | 1.00 | 2.00 | 3.00 |
| Pain | Frequent | 0 | 1.33 | 2.33 | 3.33 |
| | Almost continues | 0 | 1.66 | 2.66 | 3.66 |

| Neuropathic | Symptoms frequency Symptom into | | | | |
|---|---|---|---|---|---|
| symptoms | | Absent | Slight | Moderate | Severe |
| 2.Burning | Occasional | 0 | 1.00 | 2.00 | 3.00 |
| pain | Frequent | 0 | 1.33 | 2.33 | 3.33 |
| | Almost continues | 0 | 1.66 | 2.66 | 3.66 |

| Neuropathic Symptoms frequency Sym | | | Symptom intensity | | |
|---|---|---|---|---|---|
| symptoms | | Absent | Slight | Moderate | Severe |
| 3.Paraesthesia | Occasional | 0 | 1.00 | 2.00 | 3.00 |
| | Frequent | 0 | 1.33 | 2.33 | 3.33 |
| | Almost continues | 0 | 1.66 | 2.66 | 3.66 |

| Neuropathic | Symptoms frequency | Symptom intensity | | | |
|---|---|---|---|---|---|
| symptoms | | Absent | Slight | Moderate | Severe |
| 4.Numbness | Occasional | 0 | 1.00 | 2.00 | 3.00 |
| | Frequent | 0 | 1.33 | 2.33 | 3.33 |
| | Almost continues | 0 | 1.66 | 2.66 | 3.66 |

# 2. Neuropathy Symptom Score (NSS)

| Symptoms | |
|-------------------------------------|---|
| Burning, numbness, tingling | 2 |
| Fatigue, cramping, aching | 1 |
| None | 0 |
| Location | |
| Feet | 2 |
| Calves | 1 |
| Elsewhere | 0 |
| Timing of symptoms | |
| Nocturnal exacerbation | 2 |
| Present during day and night | 1 |
| Present during the day only | 0 |
| Symptoms wake patient up from sleep | 1 |
| Manoeuvres to reduce symptoms | |
| Walking | 2 |
| Standing | 1 |
| Sitting/Lying | 0 |
| NSS score | |

## 3. The revised version of Diabetes Quality of Life (RV-DQoL) questionnaire

Please read each statement carefully and mark the number that best suits you.

| Satisfaction Domain | Very satisfied | Moderately satisfied | Neither<br>satisfied nor<br>dissatisfied | Moderately<br>dissatisfied | Very<br>dissatisfied |
|---|---|---|---|---|---|
| 13. How satisfied are you with the amount of time it takes to manage your diabetes? | 1 | 2 | 3 | 4 | 5 |
| 14. How satisfied are you with the amount of time you spend getting checkups? | 1 | 2 | 3 | 4 | 5 |
| 15. How satisfied are you with the time it takes to determine your sugar level? | 1 | 2 | 3 | 4 | 5 |
| 16. How satisfied are you with your current treatment? | 1 | 2 | 3 | 4 | 5 |

| 17. How satisfied are you with your knowledge about your diabetes? | 1 | 2 | 3 | 4 | 5 |
|---|---|---|---|---|---|
| 18. How satisfied are you with life in general? | 1 | 2 | 3 | 4 | 5 |

| Impact Domain | Never | Sometimes | Often | Frequently | Always |
|---|---|---|---|---|---|
| 9. How often do you feel pain associated with the treatment for your diabetes? | 1 | 2 | 3 | 4 | 5 |
| 10. How often do you feel physically ill? | 1 | 2 | 3 | 4 | 5 |
| 11. How often does your diabetes interfere with your family life? | 1 | 2 | 3 | 4 | 5 |
| 12. How often do you find your diabetes limiting your social relationships and friendships? | 1 | 2 | 3 | 4 | 5 |

| W | Vorry Domain | Never | Sometimes | Often | Frequently | Always |
|---|---|---|---|---|---|---|
| 7. | How often do you worry about whether you will pass out? | 1 | 2 | 3 | 4 | 5 |
| 8. | How often do you worry that your body looks different because you have diabetes? | 1 | 2 | 3 | 4 | 5 |
| 9. | How often do your worry that you will get complications from your diabetes? | 1 | 2 | 3 | 4 | 5 |

### 4. Clinical Data

| 1 | Body mass index (BMI) | | | kg/m <sup>2</sup> |
|---|---|---|---|---|
| | Weight: | | | 8 |
| | Height: | | | |
| 2 | Blood Pressure | | | |
| | Diood i ressure | | | mmHg |
| <u> </u> | | | ı | |
| 5. | Blood test results at the | 3 <sup>rd</sup> visit | | |
| | lood Test | | esult | |
| FF | BS (mmol/L) | | | |
| | balc (%) | | | |
| | C (mmol/L) | | | |
| - | | | | |
| - | DL (mmol/L) | | | |
| | DL (mmol/L) | | | |
| | G (mmol/L) | | | |
| Cı | reatinine | | | |
| Uı | rea | | | |
| A | ST | | | |
| A | LT | | | |
| - | LP | | | |
| 6. | Medication side effect: ☐ Yes State if applicable: | □No | | |
| 7. | i | | | |
| 8. | If you do not yake medicine? ☐ Once a week | cine every d | ay, state how of | ten in a week you do not take |

| | □2-3 times a week |
|----|-------------------------------------------------------|
| | ☐ More than 3 times a week |
| 9. | State the reason you are not taking medicine ☐ Forgot |
| | ☐ Side effects |
| | ☐ Others reasons - Specify |